CLINICAL TRIAL: NCT07258667
Title: NICOLHON - Pilot Study of the Efficacy of Nicotinamide (Vitamin B3) in Leber's Hereditary Optic Neuropathy
Brief Title: Pilot Study of the Efficacy of Nicotinamide (Vitamin B3) in Leber's Hereditary Optic Neuropathy
Acronym: NICOLHON
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 49RC25_0169; 2025-524343-13-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Leber Hereditary Optic Neuropathy (LHON); Leber's Hereditary Optic Neuropathy (LHON); Mitochondrial Disease; Optic Nerve Disease
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber; Mitochondrial Diseases; Optic Nerve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nicotinamide (Experimental)
  Interventions: Drug: Nicotinamide treatment

INTERVENTIONS:
Drug: Nicotinamide treatment — All participants receive nicotinamide (vitamin B3) at a dose of 2 grams per day for 12 months. This is an open-label, single-arm study where each patient serves as their own control. Outcomes will be compared longitudinally to baseline measurements.

SUMMARY:
Leber Hereditary Optic Neuropathy (LHON) is a rare genetic disease that causes sudden and severe vision loss, usually in young adults. It is linked to mutations in mitochondrial DNA that impair energy production in retinal ganglion cells, leading to degeneration of the optic nerve. Currently, treatment options are very limited and often ineffective. Recent research has shown that patients with LHON have lower levels of nicotinamide (vitamin B3), a key molecule for mitochondrial energy metabolism. Nicotinamide is a precursor of NAD, an essential cofactor for cellular energy production. Experimental studies and clinical trials in related optic nerve diseases suggest that nicotinamide may protect retinal ganglion cells. Our hypothesis is that supplementation with high-dose nicotinamide could restore NAD levels, support mitochondrial activity, and help preserve or improve vision in LHON. This pilot study will evaluate the effectiveness and safety of oral nicotinamide (2 grams per day for 12 months) in patients who developed LHON within the past 18 months and carry one of the two most severe mutations (m.11778G>A or m.3460G>A). The main goal is to measure changes in visual acuity over time using standardized eye charts. Secondary objectives include assessing visual fields, retinal structure by optical coherence tomography (OCT), blood nicotinamide levels, and quality of life. Liver function will be monitored to ensure safety. If this study shows promising results, it could pave the way for a larger randomized trial and ultimately offer a new therapeutic option.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16 years or older.
* Diagnosis of Leber Hereditary Optic Neuropathy (LHON) due to a confirmed mitochondrial DNA mutation m.11778G>A or m.3460G>A.
* Onset of LHON symptoms less than 18 months before inclusion.
* Naïve to nicotinamide treatment for at least 3 months prior to inclusion.
* Able to take oral medication and comply with study procedures.
* Affiliated with or beneficiary of a social security system.
* Signed informed consent (or parental consent for minors; assent for minors when applicable).

Exclusion Criteria:

* Asymptomatic carriers of m.11778G>A or m.3460G>A mutations (no clinical LHON).
* LHON due to other mitochondrial DNA mutations or nuclear DNA mutations.
* LHON onset more than 18 months before inclusion.
* Current or recent treatment with idebenone (within 3 months).
* Severe associated ophthalmologic disease (e.g., advanced glaucoma, retinal pathology).
* Patients treated with gene therapy.
* Elevated liver enzymes (ASAT and/or ALAT > 2× upper normal limit) at screening or within 2 months prior to inclusion.
* Pregnant, breastfeeding, or postpartum women.
* Known contraindication to nicotinamide or allergy/intolerance to lactose or galactose.
* Persons deprived of liberty by judicial or administrative decision.
* Subjects under legal protection or psychiatric care under constraint.
* Unable to provide informed consent.
* Participation in another interventional study affecting LHON management.
* Any condition that, in the investigator's judgment, could compromise patient safety or study integrity.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of administering 2 grams per day of nicotinamide for 12 months in patients who have developed NOHL due to an m.11778G>A or m.3460G>A mutation within the last 18 months. | inclusion, 3 months, 6 months, 9 months, and 12 months
  Evaluation by the change in corrected distance visual acuity measured eye by eye on an ETDRS (Early Treatment Diabetic Retinopathy Study) scale over the entire follow-up period.

SECONDARY OUTCOMES:
The effectiveness of treatment on the progression of corrected distance visual acuity | 12 months
  Measurement eye by eye using the ETDRS scale, taking the nadir (lowest visual acuity reached a few weeks after the onset of NOHL) as the reference value.
The effectiveness of treatment on the evolution of corrected distance visual acuity | inclusion, 3 months, 6 months, 9 months and 12 months
  Measurement eye by eye on a Monoyer scale. Reading capital letters at a distance of 5 meters. Each line on the wall-mounted optometric chart corresponds to 1/10 of visual acuity.The dimensions of the letters are such that they measure 5 times the distance of discrimination corresponding to the measured visual acuity.0.4/10 is low visual acuity and 20/10 is good visual acuity.
The effectiveness of treatment on the evolution of corrected near visual acuity | inclusion, 3 months, 6 months, 9 months and 12 months
  Measurement eye by eye on a Parinaud scale; different sizes of typeface is placed at 33cm. The test consists of a text whose paragraphs are written in decreasing font sizes. The result is expressed in P (P1.5 to P50). The higher the P, the poorer the acuity.
The effectiveness of treatment on the evolution of Campimetric deficits | inclusion, 3 months, 6 months, 9 months and 12 months
  The average and corrected average deviation measured in STAT 30 on an automated visual field
The effectiveness of treatment on the evolution of the appearance of visual field | inclusion, 3 months, 6 months, 9 months and 12 months
  By the Goldman-type manual
The effectiveness of treatment on the evolution of optic nerve fiber layer (RNFL) thickness | inclusion, 3 months, 6 months, 9 months and 12 months
  Measurement by optical coherence tomography (OCT)
The effectiveness of treatment on the evolution of retinal ganglion cell complex (GCC) | inclusion, 3 months, 6 months, 9 months and 12 months
  Measurement by optical coherence tomography (OCT)
The effectiveness of treatment on the evolution of Patients' quality of life | inclusion and 12 months
  NEI VFQ 25 questionnaire. Individual scores are recoded and transformed on a scale of 0 to 100, where 100 represents the best possible functioning and 0 the worst. An average score is calculated for each of the 12 subscales.
Biological efficacy of treatment | 3 and 12 months
  Nicotinamide levels in patients' blood
Treatment tolerance on Hepatic toxicity | Inclusion, 3 months, 6 months, 9 months, 12 months
  Transaminase levels
Treatment tolerance in the macula | Inclusion, 3 months, 6 months, 9 months, 12 months
  Measurement by optical coherence tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared at a later date upon request (e.g., the CRF to allow a collaborator to select the data they wish to access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the study investigator, based on a protocol provided by the requester, after verification of the obtaining of regulatory approvals, including the favorable opinion of an ethics committee. Supporting information
Supporting Information: Study Protocol
Time Frame: The data will be shared after signing a negotiated data transfer agreement ( data access agreement), for the duration specified in the agreement
Access Criteria: The data will be made available via secure transfer (sharing platform approved by the university hospital: BlueFiles or Oodrive).